### The UNIVERSITY OF CHICAGO

The Division of the Biological Sciences • The University of Chicago Medical Center

# CONSENT/AUTHORIZATION BY SUBJECT FOR PARTICIPATION IN A RESEARCH PROTOCOL

| Protocol Number: 15-1115 | Name of Subject: |
|--------------------------|-------------------------|
| | Medical History Number: |

## **STUDY TITLE**:

"A Double-Blind, Placebo-Controlled Study of Vortioxetine in the Treatment of Binge Eating Disorder"

Doctors Directing Research: Dr. Jon Grant & Dr. Royce Lee

Address: 5841 S. Maryland Ave, Chicago, IL 60637

**Telephone Number**: 773-834-1325

You are being asked to participate in a research study. A member of the research team will explain what is involved in this study and how it will affect you. This consent form describes the study procedures, the risks and benefits of participation, as well as how your confidentiality will be maintained. Please take your time to ask questions and feel comfortable making a decision whether to participate or not. This process is called informed consent. If you decide to participate in this study, you will be asked to sign this form.

#### WHY IS THIS STUDY BEING DONE?

The aim of the present study is to examine the efficacy and safety of vortioxetine vs placebo (a pill that contains no medicine) in adults with Binge Eating Disorder. This research is being done because the researchers want to find out if vortioxetine works in reducing the symptoms of Binge Eating disorder significantly more than a placebo. The study drug, vortioxetine, is an experimental drug that has been approved by the FDA for the treatment of Major Depressive Disorder but is not approved to treat Binge Eating Disorder. The use of vortioxetine in this study is therefore considered experimental.

## HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

About 80 people will take part in this study at the University of Chicago.

## WHAT IS INVOLVED IN THE STUDY?

Based on your telephone screening, you may be eligible for this study. We have asked you to come in for a screening visit. After signing this consent form, you will undergo the following to determine if you are eligible:

- A review of your medical history, a review of medications you have taken and any past treatments for binge eating will be completed.
- You will undergo a psychiatric interview, which entails a structured clinical interview of psychiatric disorders with a research team member.

- You will be asked to give a urine sample that will be tested for drug use. This test must be negative for you to participate in the study.
- If you are a female capable of having a child, you will be given a urine pregnancy test to ensure that you are not pregnant at the time of study entry. This test must be negative for you to participate in the study, and you also must be using appropriate contraceptives during the course of the study. Additionally, you must not be breastfeeding.

Based on the result of this interview, we will determine if you qualify the study. If so, we will ask you to complete the following Baseline Visit procedures at this same visit:

- You will have a physical exam and your sitting and standing blood pressure, pulse, temperature, weight and height will be recorded.
- You will be asked if you are willing to provide an optional blood sample (3 teaspoons) to measure blood glucose level (blood sugar) to check for diabetes. If you consent, your blood will be drawn one time. If you do not consent to having your blood drawn, you are still eligible to participate in this study.

I agree to have an optional blood draw to measure my blood glucose level to check for diabetes.

| YES | NO | |
|-----|----|-------------------|
| | | Initials and date |

- An Electrocardiogram (EKG- an electrical tracing of your heart) will be obtained to check your heart activity if your medical history suggests cardiac problems.
- You will be asked about how you are feeling and if you have recently started taking any new medications or had any other changes to other medications recently.
- You will be asked to complete several forms related to binge eating, including both self-report and clinician administered inventories.
- You will also be asked to complete questionnaires about anxiety, depression, mood and other behaviors.
- You will be asked to complete a series of computer tasks measuring attention and impulsivity.
- You will be asked to complete a binge eating diary, which includes writing down the
  time of day the binge occurred, the number of binges, the time spent on the binge, the
  estimated calories of each binge, and what you ate during the binge. You will be
  given information sheets where you can keep track of this information and we will
  review the diary at each visit.
- You will receive the study drug you have been randomly assigned to for the study. The study drug is provided in the form of a pill which you take by mouth.

This baseline visit will require approximately 2-3 hours.

Study Drug Administration

Following the baseline visit, the study drug administration phase will begin. You will be randomly assigned to receive either the active study drug vortioxetine or the placebo. The placebo does not contain any active drug. The random assignment is based on a 50/50 chance, like flipping a coin. Neither the study personnel nor you will know whether you are taking vortioxetine or the placebo. This is what is meant by "blinding." The study will last up to 13-weeks and involves up to 9 study visits, including the baseline visit. You will take your assigned study drug for the duration of the 13 weeks.

You will start by taking 10mg of vortioxetine or placebo for the first 7 days of the study. After the first 7 days, you will go up to 20mg of the vortioxetine (or remain on placebo). You will remain on 20mg of vortioxetine or placebo until the last week of the study (for a total of 11 weeks). Then you will taper off of the study drug by going down on dose to 10mg during the last 7 days of the study.

The study doctor will discuss the next study visit scheduling with you during each of your current visits.

For the first 3 visits (Visit 1, Visit 2, and Visit 3), visits will be scheduled one week apart. Visits 4-8 will be scheduled two weeks apart.

During Visits 2-7, the following will occur:

- Your weight and vital signs will be checked.
- You will be given the study drug or placebo.
- You will be asked to complete several questionnaires to assess binge eating behavior and mood since the last visit.
- These visits will take approximately 30 minutes to one hour each.

Visit 8 will be scheduled two weeks after Visit 7, and the following will occur:

- You will have a physical exam and your sitting and standing blood pressure, pulse, temperature, weight and height will be recorded.
- You will be asked about how you are feeling and if you have started taking any new medications or had any other changes to other medications you may be taking since your last visit.
- You will be asked to complete the same forms administered during the first visit, including the cognitive tasks on the computer.

The final visit (Visit 9) will be scheduled one week after Visit 8 and we will ask about any problems or side effects you might be experiencing.

During this study, Dr. Grant and his research team will collect information about you for the purposes of this research. This information will include the following: your name, contact information, social security number (for payment purposes), basic demographic information (such as your age, gender, and race), relationship status, sexual orientation, family and other history, medical and medication history, and responses from questionnaires. This information is being collected so that we are able to later evaluate your information and other participants' to find correlations between certain

characteristics and mood and treatment outcomes. This information is also being collected so that we are able to compare those results to different outcomes and to other participants. All of the data collected will be completely confidential.

## **HOW LONG WILL I BE IN THE STUDY?**

We think you will be in the study for about 13 weeks. There is no long-term follow-up in the study after you stop the study drug.

Dr. Grant may decide to take you off of the study without your consent if:

- You are unable to meet the requirements of the study;
- Your medical condition changes;
- The study drug is no longer available;
- New information becomes available that indicates that participation in this study is not in your best interest; or
- If the study is stopped.

# WHAT ARE THE RISKS OF THE STUDY?

You may experience side-effects while taking the drug used in this study. Your condition may remain the same or worsen if this treatment does not work for you.

The most common side effects associated with vortioxetine include (percentages are the expected frequency):

- nausea (30%)
- diarrhea (7%)
- constipation (6%)
- vomiting (6%)
- dry mouth (8%)
- flatulence (1%)
- dizziness (9%)
- sexual dysfunction (5% in males, 2% in females)

Vortioxetine and other similar drugs may increase suicidal thoughts or actions in some children, teenagers, or young adults within the first few months of treatment or when the dose is changed. Notify study staff immediately if you experience these symptoms.

There may be risks to taking vortioxetine that are not now known. If new information becomes available which could influence your willingness to continue, this new information will be discussed with you.

The use of drugs that modulate serotonin, including vortioxetine, may increase the risk of bleeding events. Using aspirin, nonsteroidal anti-inflammatory drugs (NSAIDS), warfarin, and other anticoagulants along with vortioxetine may further increase this risk. If you have questions about what medications you can or cannot take with the study drug, feel free to ask Dr. Grant or the research staff at any time.

There have been reports of serious, sometimes **fatal**, reactions between drugs that modulate serotonin, such as vortioxetine, and monoamine oxidase inhibitors (MAOI) (another type of drug commonly used for depression). Therefore, it is recommended that vortioxetine should not be used in combination with an MAOI, or within 14 days of stopping treatment with an MAOI. Similarly, at least 14 days should be allowed after stopping vortioxetine before starting an MAOI. Again if you have questions about this, please ask Dr. Grant.

If you consent to having your blood drawn, the needle stick may cause discomfort, pain, burning sensation, or bruising.

If you are asked to get an EKG, you may have some discomfort when the electrodes (soft patches attached using adhesive tape) are removed from your chest and limbs. There is a possibility you could develop a minor rash when the electrodes were placed. This rash should go away without treatment.

It is possible that some of the questions may cause discomfort or mental stress, such as "do you feel down or sad?" and specific questions that involve your binge eating habits. If that should happen, we would be happy to talk about any thoughts or problems you may have. The study doctor may remove subjects from this study who have suicidal thoughts. In such a case, the study doctor may refer you for additional help.

## ARE THERE ANY BENEFITS TO TAKING PART IN THE STUDY?

If you agree to take part in this study, there may or may not be direct medical benefit to you for your binge eating behavior. We hope the information learned from this study will benefit other individuals with binge eating disorder in the future.

# WHAT OTHER OPTIONS ARE THERE?

Instead of being in this study, you have these options:

- Receive standard of care medication given for your condition, such as Vyvanse (lisdexamfetamine dimesylate)
- Receive psychotherapy
- No treatment and/or therapy

There are a select number of treatment options which have been found to be helpful for the treatment of binge eating disorder. Dr. Grant and his research team can provide you with information on resources in Chicago where you could potentially find other options for care.

The decision whether or not you wish to participate in this study will not affect your care at the University of Chicago Medical Center.

## WHAT ARE THE COSTS?

Clinical services provided during a clinical trial are either research-related or related to usual medical care. Research-related services are done to complete the research and the costs are not the responsibility of you or your insurance.

The costs that are considered research-related for this study include the following: all vortioxetine/placebo for the duration of the study, all visits with the study team (including Dr. Grant or Dr. Lee), pregnancy tests, urine drug tests, physical exams, blood draws, EKG, and psychiatric evaluations.

Usual medical care costs include any and all services that are considered medically necessary for your disease, such as medications or treatments. The cost of this usual, ongoing medical care will be the responsibility of you or your insurance, and may include deductibles and co-payments. Similarly, this care will be subject to all the same requirements and restrictions of your insurance. Once the study has concluded, the continuation of care from a mental health provider will be the responsibility of you and/or your insurance. This would include the cost of vortioxetine, if you wish to continue taking one of them after your participation in the study has ended.

If you suffer an unanticipated injury as a direct result of this research and require emergency medical treatment, treatment will be provided at the University of Chicago Medical Center at no cost to you. You must notify Dr. Grant as promptly as possible after your injury in order to receive this care. An injury is "unanticipated" if it is not one of the known effects of vortioxetine, and is not the result of your disease or condition. The costs of any non-emergency care for such an injury will be billed to you or your insurance in the ordinary manner. If you think that you have suffered a research related injury, you must let Dr. Grant know right away.

### WILL I BE PAID FOR MY PARTICIPATION?

For participation in this study you will receive \$20 per visit. The total amount you could receive for this study is \$180 if you complete all nine study visits. All payment for your participation will be provided in the form of cash after every visit. You will also be compensated for your travel in the form of a parking voucher or bus voucher, which you will receive at the conclusion of each visit.

The policies at the University of Chicago may require that you to complete a tax form in order to receive compensation. If this is the case, we will be collecting personal information about you including your name, address, and social security number.

## WHAT ABOUT CONFIDENTIALITY?

Study records that identify you will be kept confidential. All records will be kept in a secure office in a locked cabinet of the Psychiatry Department at the University of Chicago. Only study staff will have access to study records. The data collected in this study will be used for the purpose described in the form. By signing this form, you are allowing the research team access to your medical records, which include Protected Health Information. Protected Health Information (PHI) consists of any health information that is collected about you, which could include your medical history and new information collected as a result of this study. The research team includes the individuals listed on this consent form and other personnel involved in this study at the University of Chicago.

As part of the study, Dr. Grant and his research team will report the results of your study-related procedures and tests explained above to Takeda Pharmaceuticals. These include any serious adverse effects that may occur during the course of the study. This information is being sent because the sponsor needs to be informed of any serious problems that may occur with the study drug for monitoring and drug labeling purposes. The study sponsor or their representatives, including monitoring agencies, may also review your medical record. Please note that these individuals may share your health information with someone else.

Your records may be reviewed by federal agencies whose responsibility is to protect human subjects in research including the Food and Drug Administration (FDA) and Office of Human Research Protections (OHRP). In addition, representatives of the University of Chicago, including the Institutional Review Board, a committee that oversees the research at the University of Chicago, may also view the records of the research. If your research record is reviewed by any of these groups, they may also need to review your entire medical record.

If health information is shared outside the University of Chicago, the same laws that the University of Chicago must obey may not protect your health information.

During your participation in this study, you will have access to your medical record. Dr. Jon Grant is not required to release to you research information that is not part of your medical record.

This consent form will be kept by the research team for at least six years. The study results will be kept in your research record and be used by the research team indefinitely. At the time of study completion, either the research information not already in your medical record will be destroyed or information identifying you will be removed from study results. Any research information in your medical record will be kept indefinitely.

Data from this study may be used in medical publications or presentations. Your name and other identifying information will be removed before this data is used. If we wish to use identifying information in publications, we will ask for your approval at that time.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## WHAT ARE MY RIGHTS AS A PARTICIPANT?

Taking part in this study is voluntary. If you choose not to participate in this study, your care at the University of Chicago/University of Chicago Medical Center will not be affected. You may choose not to participate at any time during the study. Leaving the study will not affect your care at the University of Chicago/University of Chicago Medical Center.

If you choose to no longer be in the study and you do not want any of your future health information to be used, you must inform Dr. Grant in writing at the address on the first page. Dr. Grant may still use your information that was collected prior to your written notice.

We will tell you about significant new information that may affect your willingness to stay in this study.

You will be given a signed copy of this document. This consent form document does not have an expiration date.

# WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

You have talked to Dr. Grant about this study and you had the opportunity to ask questions concerning any and all aspects of the research. If you have further questions about the study, you may call Dr. Grant at 773-834-1325.

If you have a research related injury, you should call Dr. Grant (the study doctor) immediately at 773-834-1325.

If you have any questions concerning your rights in this research study you may contact the Institutional Review Board, which is concerned with the protection of subjects in research projects. You can reach the Committee office between 8:30 am and 5:00 pm, Monday through Friday, by calling (773) 702-6505 or by writing: University of Chicago, Institutional Review Board, 5841 S. Maryland Ave., MC7132, I-624, Chicago, IL 60637.

## **CONSENT**

#### **SUBJECT**

The research project and the procedures associated with it have been explained to me. The experimental procedures have been identified and no guarantee has been given about the possible results. I will receive a signed copy of this consent form for my records.

I agree to participate in this study. My participation is voluntary and I do not have to sign this form if I do not want to be part of this research study.

| Signature of Subject: | | |
|---|---|---|
| Date: | Time: | AM/PM (Circle) |
| PERSON OBTAINING CONSENT I have explained to the nature and purpose of the study and the risks involved. I have answered and will answer all questions to the best of my ability. I will give a signed copy of the consent form to the subject. | | |
| Signature of Person Obtaining Consent: | | |

| Date: | Time: | AM/PM (Circle) |
|---|---|---|
| INVESTIGATOR/PI<br>Signature of Investig | | |
| Date: | Time <sup>.</sup> | AM/PM (Circle) |